CLINICAL TRIAL: NCT02046356
Title: Recurrence Risk Factors of Early-Stage Hepatocellular Carcinoma After Radio Frequency Ablation: a Multi-center Prospective Case-control Study
Brief Title: Recurrence Risk Factors of Early-Stage Hepatocellular Carcinoma After Radio Frequency Ablation
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Yunhua Tan (Other)
Collaborators: Southwest Hospital, China (Other)
Responsible Party: Sponsor-Investigator, Yunhua Tan, Instructor, Southwest Hospital, China
Organization: Southwest Hospital, China (Other)
Other Study IDs: SWH-66; SouthwestH (Other: SouthwestH)
Record Dates: First submitted 2014-01-23; First posted 2014-01-27 (Estimated); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; radiofrequency ablation; Milan Criteria; recurrence; risk factor
MeSH Terms: conditions — Carcinoma, Hepatocellular; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Early-Stage HCC: Early-Stage hepatocellular carcinoma From January 2014 to January 2015, a total of 139 patients with early HCC from the First Affiliated Hospital, the Second Affiliated Hospital and the Third Affiliated Hospital of the Third Military Medical University were prospectively recruited according after MESS-RFA
  Interventions: Procedure: MESS-RFA

INTERVENTIONS:
Procedure: MESS-RFA

SUMMARY:
The aim was to investigate the efficacy of radiofrequency ablation (RFA) with a multiple-electrode switching system (MESS) in the treatment of early hepatocellular carcinoma (HCC) and to evaluate the patterns and risk factors of intrahepatic recurrence of HCC after RFA.

DETAILED DESCRIPTION:
Percutaneous RFA has become a particularly promising treatment for patients with early HCC. For HCC with a diameter less than 3cm, RFA is becoming an effective topical method for the goal of a complete cure. Although RFA is successful for small HCCs, for HCCs with a diameter larger than 3 to 5 cm, the complete ablation rate is reported to range from 61.3% to 82.5%. These results may be obsolete due to the further development of RFA techniques and instruments. For example, the use of clustered electrodes and an improved motor can provide a higher power, and the multiple-electrode switching system RFA (MESS-RFA) uses various methods to create a sufficient ablation zone, the investigators need to further update the management strategy of the RFA treatment of early HCC.

However, HCC recurrence after RFA is still a significant problem . the investigators divide the intrahepatic recurrence after RFA into local tumor progression (LTP) and intrahepatic distant recurrence (IDR); each type of recurrence has a different pathogenic mechanism and is thought to occur relatively independently . Understanding the pattern and risk factors of recurrence is very important for the development of RFA and its clinical application.

The objective of our multicenter prospective study was to evaluate the efficacy of MESS-RFA as a primary method for treating early HCC, to assess the pattern of intrahepatic recurrence according to the types of recurrence, and to determine the risk factors associated with tumor recurrence and survival.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years old
* The diameter of single tumor should be no more than 5cm, or multiple tumors(less than 3 loci) should be no more than 3cm. No large vascular invasion, no lymph nodes or extrahepatic metastases
* The Classification of patients' liver function is Child - Pugh A or B
* No serious coagulation dysfunction (prothrombin activity < 40% or platelet count < 30000 / mL).
* No refractory ascites.
* The patients can be treated with RFA in clinical
* Primary treatment by RFA should ablate the tumor(s) completely
* The patients are aware of their condition, the treatment of the HCC, and the risks associated with radiofrequency ablation therapy.
* The patients participant voluntarily and they will sign the informed consent before the radiofrequency ablation therapy.

Exclusion Criteria:

* The patients are from abroad, Hong Kong, Macao, Taiwan and other regions, who are impossible to be follow-up
* The patients who refuse to sign the informed consent
* Tumor emboli existed in main portal vein, ductus hepatics communis and(or) its primary branch, main hepatic vein and(or) inferior vena cava before operation
* Extrahepatic metastasis, lymph node metastasis
* The patients whom accept systemic chemotherapy, preoperative interventional therapy, and(or) other auxiliary treatment
* The patients with diabetes mellitus, heart disease and(or) other diseases can't tolerate radiofrequency ablation, or influence postoperative follow-up
* The existence of other type of malignant tumor before or accompanied by HCC
* Primary treatment by RFA do not ablate the tumor(s) completely
* Non-primary liver tumor, such as the liver metastatic carcinoma, cholangiocarcinoma, etc

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In-patients from three affiliated hospital of the Third Military Medical University
Sampling Method: Non-Probability Sample
Enrollment: 139 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Technical success | up to 5 years
  Complete ablation rate

SECONDARY OUTCOMES:
LTP | up to 5 years
  local tumor progression
IDR | up to 5 years
  intrahepatic distant recurrence
Overall survival | up to 5 years
  Overall survival rates
IDR-free survival | up to 5 years
  IDR-free survival rates

OTHER OUTCOMES:
RFA complications | up to 5 years
  Complication rate

CONTACTS AND LOCATIONS:
Overall Officials: Yunhua Tan, Principal Investigator — Southwest Hospital, China
Locations (1):
- Southwest hospital, Chongqing, Chongqing Municipality, China

REFERENCES:
- [Background] Shiina S, Tateishi R, Arano T, Uchino K, Enooku K, Nakagawa H, Asaoka Y, Sato T, Masuzaki R, Kondo Y, Goto T, Yoshida H, Omata M, Koike K. Radiofrequency ablation for hepatocellular carcinoma: 10-year outcome and prognostic factors. Am J Gastroenterol. 2012 Apr;107(4):569-77; quiz 578. doi: 10.1038/ajg.2011.425. Epub 2011 Dec 13. PMID 22158026
- [Background] Arii S, Yamaoka Y, Futagawa S, Inoue K, Kobayashi K, Kojiro M, Makuuchi M, Nakamura Y, Okita K, Yamada R. Results of surgical and nonsurgical treatment for small-sized hepatocellular carcinomas: a retrospective and nationwide survey in Japan. The Liver Cancer Study Group of Japan. Hepatology. 2000 Dec;32(6):1224-9. doi: 10.1053/jhep.2000.20456. PMID 11093728
- [Background] Hasegawa K, Makuuchi M, Takayama T, Kokudo N, Arii S, Okazaki M, Okita K, Omata M, Kudo M, Kojiro M, Nakanuma Y, Takayasu K, Monden M, Matsuyama Y, Ikai I. Surgical resection vs. percutaneous ablation for hepatocellular carcinoma: a preliminary report of the Japanese nationwide survey. J Hepatol. 2008 Oct;49(4):589-94. doi: 10.1016/j.jhep.2008.05.018. Epub 2008 Jun 12. PMID 18620773
- [Background] Ng KK, Poon RT, Lo CM, Yuen J, Tso WK, Fan ST. Analysis of recurrence pattern and its influence on survival outcome after radiofrequency ablation of hepatocellular carcinoma. J Gastrointest Surg. 2008 Jan;12(1):183-91. doi: 10.1007/s11605-007-0276-y. Epub 2007 Sep 15. PMID 17874276
- [Background] Lam VW, Ng KK, Chok KS, Cheung TT, Yuen J, Tung H, Tso WK, Fan ST, Poon RT. Risk factors and prognostic factors of local recurrence after radiofrequency ablation of hepatocellular carcinoma. J Am Coll Surg. 2008 Jul;207(1):20-9. doi: 10.1016/j.jamcollsurg.2008.01.020. Epub 2008 Apr 24. PMID 18589357
- [Background] Kudo M. Radiofrequency ablation for hepatocellular carcinoma: updated review in 2010. Oncology. 2010 Jul;78 Suppl 1:113-24. doi: 10.1159/000315239. Epub 2010 Jul 8. PMID 20616593
- [Background] Lee HY, Rhim H, Lee MW, Kim YS, Choi D, Park MJ, Kim YK, Kim SH, Lim HK. Early diffuse recurrence of hepatocellular carcinoma after percutaneous radiofrequency ablation: analysis of risk factors. Eur Radiol. 2013 Jan;23(1):190-7. doi: 10.1007/s00330-012-2561-8. Epub 2012 Oct 20. PMID 23085860
- [Derived] Tan Y, Wang X, Ma K, Zhang L, Li J, Chen P, Zhang B. Risk factors for the recurrence of early hepatocellular carcinoma treated by percutaneous radiofrequency ablation with a multiple-electrode switching system: a multicenter prospective study. Int J Hyperthermia. 2022;39(1):190-199. doi: 10.1080/02656736.2021.2024279. PMID 35042449
- [Derived] Tan Y, Jiang J, Wang Q, Guo S, Ma K, Bie P. Radiofrequency ablation using a multiple-electrode switching system for hepatocellular carcinoma within the Milan criteria: long-term results. Int J Hyperthermia. 2018 May;34(3):298-305. doi: 10.1080/02656736.2017.1330495. Epub 2017 May 29. PMID 28554226
- See also: Southwest Hospital,China — http://www.xnyy.cn/